CLINICAL TRIAL: NCT05270239
Title: Neurorehabilitation and Functional Recovery in Multiple Sclerosis: Assessing Two Therapeutic Strategies Using Functional Magnetic Resonance Imaging.
Brief Title: Function Magnetic Resonance Imaging to Assess Two Therapeutic Strategies in Multiple Sclerosis (NeuroRehEM).
Acronym: NeuroRehEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PID2019-106793RB-I00
Record Dates: First submitted 2022-01-31; First posted 2022-03-08 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Magnetic Resonance Imaging; Neuroplasticity; Cognitive Impairment; Virtual Reality
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working Memory Training in MS patients (Experimental): This group of patients will perform a computerized n-back training, which includes a sequence of 2-back and 3-back blocks.
  Interventions: Behavioral: N-back Cognitive Training
- Virtual Reality Training in MS patients (Experimental): This group of patients will perform a Virtual Reality "Ball Task" training. This task contains 6 trials of increasing difficulty.
  Interventions: Behavioral: Virtual Reality Motor and Cognitive Training

INTERVENTIONS:
Behavioral: N-back Cognitive Training — N-back task mainly trains working memory and information processing speed. This training lasts 10 days (1 hour per day).
  Arms: Working Memory Training in MS patients
Behavioral: Virtual Reality Motor and Cognitive Training — Virtual Reality "Ball Task" mainly trains inhibitory control, attention, working memory and motor functions. This training lasts 10 days (30 minutes per day)
  Arms: Virtual Reality Training in MS patients

SUMMARY:
Multiple sclerosis (MS) is an autoimmune disease that causes cognitive and motor disabilities and contributes to decrease patients life quality. Previous results described that there are some MS patients that showed (at least in some phases of the disease) neuroplasticity processes that are able to compensate some cognitive deficits. Moreover, neuroplasticity processes seem to be limited and related to the degree of gray matter atrophy (patients with less atrophy show grater neuroplasticity than those with higher atrophy level). The aims of this project are:

1. to study behavioral changes (post-training) induced by two different rehabilitation programs: a)cognitive training focused on exclusively enhancing working memory and b) aerobic + cognitive training aimed to enhance attention, working memory processes and motor capabilities using a virtual reality game.
2. to study neuroplasticity changes (post-training functional connectivity changes) induced by these rehabilitation programs
3. to observe the role of the atrophy in brain neuroplasticity processes.

Neuropathological status and neuroplasticity processes (studied using neuroimaging tools) as well as cognitive performance using neuropsychological tools will be assessed in a group of MS patients (with different phenotypes) at two different time points: before any training (S1) and after 10 days of training (S2). This project will be financed by the Ministerio de ciencia, innovación y universidades of the Spanish government and also have been approved by the Ethical committee of Universitat Jaume I.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis Diagnosis.

Exclusion Criteria:

* Other neurological pathologies comorbidity.
* Magnetic resonance imaging incompatibilities.
* Motor impairment degree that impede the task performance.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Correct Responses | Baseline and 10 training days after.
  Number of correct responses in both tasks (n-back computerized task and balls Virtual Reality task)
Change from baseline in Reaction Time | Baseline and 10 training days after.
  This is a primary outcome of the n-back task, which refers to the amount of time (in milliseconds) that elapse from the moment the correct stimulus appears and the correct response is given.
Change from baseline in Omissions | Baseline and 10 training days after.
  In both tasks will be assessed the number of times that a correct stimulus appear and non-response is given.
Change from baseline in Errors | Baseline and 10 training days after.
  The number of times that a distractor stimulus appears and a response is given.
Change from baseline in Functional Connectivity in resting state | Baseline and 10 training days after.
  This is a brain activity measure during resting state through functional magnetic resonance imaging. This outcome will be assessed in both studies.
  fMRI sequence: T2-weighted echoplanar imaging sequence.
Change from baseline in Functional Connectivity in task performance | Baseline and 10 training days after.
  This is a brain activity measure during a task performance through functional magnetic resonance imaging. This outcome will be assessed in Virtual Reality study.
  fMRI sequence: T2-weighted echoplanar imaging sequence.
Change from baseline in SRT-S: Selective Reminding Test (Storing) | Baseline and 10 training days after.
  A subtest of the BRB-N (The Brief Repeatable Battery of Neuropsychological Tests for MS) which measures memory storage capacity.
Change from baseline in SRT-R: Selective Reminding Test (Retrieval) | Baseline and 10 training days after.
  This subtest of the BRB-N is a measure of memory retrieval capacity.
Change from baseline in SRT-D: Selective Reminding Test (Delayed) | Baseline and 10 training days after.
  This BRB-N subtest measures the delayed memory.
Change from baseline in SPART: Spatial Recall Test | Baseline and 10 training days after.
  A subtest of the BRB-N that measures spatial memory.
Change from baseline in SPART-D: Spatial Recall Test (Delayed) | Baseline and 10 training days after.
  This BRB-N subtest measures the spatial delayed memory.
Change from baseline in SDMT: Symbol Digit Modalities Test | Baseline and 10 training days after.
  A BRB-N subtest which measures information processing speed.
Change from baseline in PASAT: Paced Auditory Serial Addition Task | Baseline and 10 training days after.
  A BRB-N subtest which measures working memory.
Change from baseline in Phonemic Fluency | Baseline and 10 training days after.
  A language measure that assesses phonemic fluency.
Change from baseline in Semantic Fluency | Baseline and 10 training days after.
  A language measure that assesses semantic fluency.
Change from baseline in Digit Span Forward | Baseline and 10 training days after.
  A subtest of the Wechsler Adult Intelligence Scale (WAIS-III) that is an attention measure.
Change from baseline in Digit Span Backward | Baseline and 10 training days after.
  A WAIS-III subtest that is a working memory measure.
Change from baseline in Letters and Numbers | Baseline and 10 training days after.
  A WAIS-III subtest that measures working memory.

SECONDARY OUTCOMES:
Total Intracranial Volume (TIV) | Baseline
  A measure of brain volumetry. MRI sequence: structural T1-weighted MPRAGE sequence.
Brain Parenchymal Fraction (BPF) | Baseline
  MRI sequence: structural T1-weighted MPRAGE sequence.
Lesion Volume in white matter tissue | Baseline
  A brain damage volumetry measure. MRI sequence: structural T1-weighted MPRAGE sequence and T2-FLAIR sequence
Cortical Lesions | Baseline
  Number of brain cortical lesions. MRI Sequence: inversion recovery MRI pulse sequence (DIR).
Cortical Thickness | Baseline
  Brain cortical thickness measure. MRI sequence: structural T1-weighted MPRAGE sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Forn, Study Director — Universitat Jaume I (Castellón, Spain); Carla Sanchis, Study Director — Universitat Jaume I (Castellón, Spain)
Locations (1):
- Universitat Jaume I (ImagoBrain Research Group), Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No
Not foreseen due to the ethics committee's privacy policy on the protection of personal data. However, upon request, radiological data could be shared.

REFERENCES:
- [Background] Baltruschat SA, Ventura-Campos N, Cruz-Gomez AJ, Belenguer A, Forn C. Gray matter atrophy is associated with functional connectivity reorganization during the Paced Auditory Serial Addition Test (PASAT) execution in Multiple Sclerosis (MS). J Neuroradiol. 2015 Jun;42(3):141-9. doi: 10.1016/j.neurad.2015.02.006. Epub 2015 Apr 6. PMID 25857687
- [Background] Cruz-Gomez AJ, Ventura-Campos N, Belenguer A, Avila C, Forn C. The link between resting-state functional connectivity and cognition in MS patients. Mult Scler. 2014 Mar;20(3):338-48. doi: 10.1177/1352458513495584. Epub 2013 Jul 4. PMID 23828871
- [Background] Mitolo M, Venneri A, Wilkinson ID, Sharrack B. Cognitive rehabilitation in multiple sclerosis: A systematic review. J Neurol Sci. 2015 Jul 15;354(1-2):1-9. doi: 10.1016/j.jns.2015.05.004. Epub 2015 May 9. PMID 25998261
- [Background] Aguirre N, Cruz-Gomez AJ, Esbri SF, Miro-Padilla A, Bueicheku E, Broseta-Torres R, Avila C, Sanchis-Segura C, Forn C. Enhanced frontoparietal connectivity in multiple sclerosis patients and healthy controls in response to an intensive computerized training focused on working memory. Mult Scler Relat Disord. 2021 Jul;52:102976. doi: 10.1016/j.msard.2021.102976. Epub 2021 Apr 24. PMID 33964569
- [Background] Sandroff BM, Wylie GR, Sutton BP, Johnson CL, DeLuca J, Motl RW. Treadmill walking exercise training and brain function in multiple sclerosis: Preliminary evidence setting the stage for a network-based approach to rehabilitation. Mult Scler J Exp Transl Clin. 2018 Feb 21;4(1):2055217318760641. doi: 10.1177/2055217318760641. eCollection 2018 Jan-Mar. PMID 29497559
- [Background] Aguirre N, Cruz-Gomez AJ, Miro-Padilla A, Bueicheku E, Broseta Torres R, Avila C, Sanchis-Segura C, Forn C. Repeated Working Memory Training Improves Task Performance and Neural Efficiency in Multiple Sclerosis Patients and Healthy Controls. Mult Scler Int. 2019 Apr 16;2019:2657902. doi: 10.1155/2019/2657902. eCollection 2019. PMID 31139470